CLINICAL TRIAL: NCT07065370
Title: Intra-Operative Modified Ventilator Mechanical Power as a Predictor of Postoperative Hypoxemia In Laparoscopic Bariatric Surgeries
Brief Title: Intra-Operative Modified Ventilator Mechanical Power in Laparoscopic Bariatric Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Ahmed Elbradey, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 36241/12/22
Record Dates: First submitted 2025-06-26; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2022-11

CONDITIONS: Laparoscopic Bariatric Surgeries; Hypoxemia; Obese Patients
Keywords: mechanical power; hypoxemia; morbid obese patients; laparoscopic bariatric surgeries
MeSH Terms: conditions — Hypoxia | interventions — Tidal Volume

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patient of this group received volume-controlled ventilation with tidal volume 6-8ml/kg (predicted body weight) with respiratory rate 12-14 cycle/minute.
  Interventions: Device: Group I ( volume-controlled ventilation with tidal volume 6-8ml/kg (predicted body weight) with respiratory rate 12-14 cycle/minute.
- Group II (Experimental): Patient of this group received volume-controlled ventilation with tidal volume 6-8ml/kg (predicted body weight) with respiratory rate 18-20 cycle/minute
  Interventions: Device: Group II: (volume-controlled ventilation with tidal volume 6-8ml/kg )

INTERVENTIONS:
Device: Group I ( volume-controlled ventilation with tidal volume 6-8ml/kg (predicted body weight) with respiratory rate 12-14 cycle/minute. — Volume-controlled ventilation with tidal volume 6-8ml/kg (predicted body weight) with respiratory rate 12-14 cycle/minute.
  Arms: Group I
Device: Group II: (volume-controlled ventilation with tidal volume 6-8ml/kg ) — group received volume-controlled ventilation with tidal volume 6-8ml/kg predicted body weight with respiratory rate 18-20 cycle/minute
  Arms: Group II

SUMMARY:
To compare the effects of two levels of mechanical power on the incidence of post-operative hypoxemia in morbid obese patients undergoing laparoscopic bariatric surgeries.

Primary outcome: Incidence of postoperative hypoxemia within the first 24 hour after surgery.

DETAILED DESCRIPTION:
Postoperative pulmonary complications are estimated to occur in more than 30% of patients after major surgery and are associated with increased morbidity, mortality and healthcare costs. Therefore, it is desirable to identify potentially modifiable factors that may be associated with an increased risk of Postoperative pulmonary complications. A high tidal volume, a high driving pressure, and also a high flow and a high respiratory rate can induce lung injury. Changing one of these variables could inadvertently affect the other three variables .

Previous studies have focused on intraoperative lung-protective ventilation to prevent Postoperative pulmonary complications but have yielded equivocal results: the combination of lowering tidal volume and applying positive end-expiratory pressure, which resulted in lower driving pressures, improved postoperative pulmonary function and reduced major postoperative adverse events. Trials investigating single interventions were, however, nonconfirmatory: a single-center randomized controlled trial failed to demonstrate an effect of low (6 ml/kg) versus high tidal volumes (10 ml/kg) in patients undergoing surgery, .While tidal volume was the only randomized variable in these studies, there was an associated increase in respiratory rate, potentially offsetting the beneficial effect of lowering tidal volume. This illustrates the need for a unifying concept that integrates the effects of changes in multiple parameters when adjusting mechanical ventilation to reduce perioperative ventilator-induced lung injury .

Recently, it has been proposed that the extent of the ventilator-induced lung injury may relate to the amount of energy transferred from the ventilator to the lungs, a concept referred to as 'mechanical power . Measurement of mechanical power is determined by a combination of factors including tidal volume, inspiratory pressure, respiratory rate and inspiratory flow rate, all of which determine the amount of energy generated during mechanical ventilation.

Previous studies have demonstrated that mechanical power is associated with increased mortality in intensive care unit patients with and without Acute Respiratory Distress Syndrome . The effects of the intraoperative mechanical power on the occurrence of Postoperative pulmonary complications in abdominal surgery have not yet been investigated thoroughly. In our study, we hypothesized that decrease mechanical power of ventilator would decrease Postoperative pulmonary complications in patients undergoing laparoscopic bariatric surgery.

The purpose of the study to compare the effects of two levels of mechanical power on the incidence of post-operative hypoxemia in morbid obese patients undergoing laparoscopic bariatric surgeries

ELIGIBILITY:
Inclusion Criteria:

* Age 21-60 years
* American society of anesthesiology physical status III
* Body mass index ≥ 40 kg/m2 undergoing laparoscopic bariatric surgery.

Exclusion Criteria:

* Uncontrolled respiratory morbidity such as sever bronchial asthma or chronic obstructive pulmonary disease.
* Patients with valvular or ischemic heart diseases, or uncontrolled hypertension
* Patients with hepatic dysfunction or renal or endocrine disorders,
* Patients with history of cerebrovascular disease or uncontrolled Diabetes mellitus.
* Previous lung surgery
* Pregnant
* Patients with neuromuscular diseases

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoxemia | 24 hours postoperative

SECONDARY OUTCOMES:
Correlation between the intraoperative mechanical power and postoperative hypoxemia | 24 hours postoperative
  Pearson correlation test was used to assess Correlation between the intraoperative mechanical power and incidence of postoperative hypoxemia

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elbradey, Resident, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF